CLINICAL TRIAL: NCT01629433
Title: PHASE IV STUDY ON THE EFFECTS OF ONABOTULINUMTOXINA INTRADETRUSORIAL INJECTIONS ON BLADDER EXPRESSION OF NGF, TRKA, P75 AND TRPV1 IN PATIENTS WITH DETRUSOR OVERACTIVITY
Brief Title: Onabotulinumtoxina Intradetrusorial Injections and NGF Expression
Acronym: Onab/A-NGF
Status: Completed | Type: Observational
Sponsor: University Of Perugia (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Antonella Giannantoni, ASSOCIATE PROFESSOR OF UROLOGY, University Of Perugia
Other Study IDs: onabotulinumatoxin and NGF
Record Dates: First submitted 2012-06-20; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Overactive Detrusor; Detrusor Hyperreflexia of Bladder
Keywords: idiopathic detrusor overactivity; neurogenic dysfunction; onabotulinumtoxinA
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder biopsy specimens obtained from the postero-lateral wall of the bladder with cold cup resection. Deep bladder wall biopsy including urothelium and smooth muscle were performed. No biopsies were taken from the bladder neck or the trigone.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- botulinum A toxin: 18 patients with neurogenic DO and 7 with idiopathic DO All the patients had overactive bladder (OAB) symptoms and DO refractory to conventional anticholinergics.

SUMMARY:
In the last years, botulinum toxin type A (onab/A) has been increasingly used as a treatment option for overactive bladder symptoms in patients affected by either neurogenic and idiopathic detrusor overactivity (DO). How onab/A injected into the detrusor muscle improves overactive bladder symptoms in neurologic patients has been only partially investigated.Some evidence suggested that the neurotoxin probably reduces detrusor muscle contraction blocking detrusor muscle cholinergic innervation. However, recent experimental observations indicated that onab/A determines more complex effects on bladder activity acting on afferent innervations as well as on the efferent one. Only few experimental studies have investigated the activity of onab/A on bladder afferent nervous transmission. Experimental studies in animals showed that Nerve Growth Factor (NGF) elicits increased sensation, urgency and DO. Although there are some evidence on the ability of onab/A to improve DO and to reduce bladder and urinary content of NGF, how onab/A influences NGF expression and the expression of TrKa, p75 and TRPV1 receptors is still unclear. The hypothesis is that onab/A reduces NGF bladder tissue levels and in the same time it modulates the gene expression of NGF associated receptors (TrkA, p75 and TRPV1).

DETAILED DESCRIPTION:
NGF has been suggested to modulate neurotransmitters' release, induces synaptic reorganization and influences neuronal excitability acting on Trk/A and p75 associated receptors. Moreover, recent observations indicated that NGF-induced DO and noxious input depend on the interaction of NGF with TRPV1, that is over-expressed in overactive bladders and interstitial cystitis/painful bladder syndrome. From a clinical point of view, a decrease in urinary NGF levels has been detected in patients with DO treated with onab/A. Although there are some evidence on the ability of onab/A to improve DO and to reduce bladder and urinary content of NGF, how onab/A influences NGF expression and the expression of TrKa, p75 and TRPV1 receptors is still unclear.

ELIGIBILITY:
Inclusion Criteria:

Patients affected by refractory overactive bladder (OAB) symptoms and detrusor overactivity (idiopathic and neurogenic DO) refractory to conventional anticholinergics (at least 3 antimuscarinic agents -- tolterodine, oxybutynin and solifenacin -- each taken for at least 1 month).

Exclusion Criteria:

* OAB symptoms due to bladder outlet obstruction because of urogenital prolapse in females and benign prostatic hyperplasia in males,
* recurrent urinary tract infections,
* cognitive impairment,
* pregnancy,
* anticoagulant therapy,
* psychoactive agents modulating bladder function (venlafaxine, amitriptyline), aminoglycosides, and other drugs thought to interfere with bladder function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We consecutively enrolled 18 patients with neurogenic DO (8 patients with spinal cord injury: 7 men and 1 women, mean age: 46±2 yrs, disease duration 6.25±1 yrs; 10 patients with suprapontine bilateral lesions: 4 men and 6 women, mean age: 55±4 yrs, disease duration 6.6±1.49 yrs ) and 7 with idiopathic DO (3 men and 4 female, mean age: 53±5 yrs, disease duration 7.1±1.53 yrs). All the patients had overactive bladder (OAB) symptoms and DO refractory to conventional anticholinergics (at least 3 antimuscarinic agents -- tolterodine, oxybutynin and solifenacin -- each taken for at least 1 month). Anticholinergics were discontinued one month before entry into the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
to investigate onab/A- induced changes on gene expression of NGF, TRPV1, TrkA and p75 in bladder wall tissue of patients with neurogenic and idiopathic DO.
  All patients underwent cystoscopy with bladder wall biopsy specimens. After undergoing cystoscopy with bladder sampling patients underwent onab/A intradetrusorial injections. Patients were injected with 100 or 300 onab/A U according to the type of DO. Urodynamic studies and cystoscopies with bladder sampling were repeated 1 month later. NGF and neuroreceptors (TrkA, TRPV1, p75)gene expression have been measured with Real Time Polymerase Chain reaction. NGF bladder tissue content (protein) has been added into evaluation and measured with ELISA.

SECONDARY OUTCOMES:
To evaluate urodynamic improvements
  Improvement in uninhibited detrusor contractions' maximum pressure (cmh20).
To investigate urodynamic improvements.
  Improvement in uninhibited detrusor contractions' first volume (ml)
To investigate urodynamic improvements.
  Improvement in maximum cystometric capacity (ml).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Perugia, Dept. of Urology and Andrology, Perugia, Italy, Italy